CLINICAL TRIAL: NCT02701270
Title: Randomised, Single-blinded, Controlled, Crossover and Acute Clinical Intervention to Assess the Effect of Three Fibres on Glycaemic and Insulinaemic Responses in Healthy Adult Volunteers
Brief Title: Effect of Three Fibres on Glycaemic and Insulinaemic Responses in Healthy Adult Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 111031-DP-2015-06-26
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: Glycemic Index; Dietary Fiber
MeSH Terms: interventions — polydextrose; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental Dietary Fibre 1 (Experimental)
  Interventions: Dietary Supplement: Experimental Dietary Fibre 1
- Experimental Dietary Fibre 2 (Experimental)
  Interventions: Dietary Supplement: Experimental Dietary Fibre 2
- Polydextrose (Active Comparator)
  Interventions: Dietary Supplement: Polydextrose
- Dextrose control (Active Comparator)
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Dietary Supplement: Experimental Dietary Fibre 1 — 22.17 g of product diluted in 250 ml of water taken once orally.
  Arms: Experimental Dietary Fibre 1
Dietary Supplement: Experimental Dietary Fibre 2 — 21.84 g of product diluted in 250 ml of water taken once orally.
  Arms: Experimental Dietary Fibre 2
Dietary Supplement: Polydextrose — 21.48 g of product diluted in 250 ml of water taken once orally.
  Arms: Polydextrose
Dietary Supplement: Dextrose — 23.89 g of dextrose diluted in 250 ml of water taken once orally.
  Arms: Dextrose control

SUMMARY:
The purpose of this study is to determine whether DuPont Experimental Dietary Fibre products 1 and 2 are digested using glycaemic and insulinaemic response as markers.

DETAILED DESCRIPTION:
DuPont Experimental Dietary Fibre products 1 and 2 glycaemic and insulinaemic response will be compared against that of polydextrose and dextrose when given to adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-27 kg/m2.
* Self-diagnosed as healthy at the time of recruitment, confirmed by medical questionnaire: no reported current or previous metabolic diseases or chronic gastrointestinal disorders.
* No blood donations during the study.
* Reported intense sporting activities < 10hr/w.
* Reported alcohol consumption ≤21 units/w (female volunteers) or ≤28 units/w (male volunteers).
* Feasibility to give blood sample as per study protocol.
* Informed consent signed

Exclusion Criteria:

* Dislike, allergy or intolerance to test products.
* Fasting blood glucose levels <4.4 or >6.1.
* Volunteer has any health conditions that would prevent him/her from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the Principal Investigator.
* Volunteer with history of diabetes and high blood pressure.
* Having consumed anything apart from plain water in the twelve hours prior to the first test day.
* Volunteer and/or immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the clinical research organization.
* Reported lactating (or lactating < 6 weeks ago), pregnant (or pregnant < 3 months ago) or wish to become pregnant during the study.
* Reported participation in another biomedical trial 1 month before the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Leatherhead Food Research, Leatherhead, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasselwander O, DiCosimo R, You Z, Cheng Q, Rothman SC, Suwannakham S, Baer ZC, Roesch BM, Ruebling-Jass KD, Lai JP, Hurteau RE, Marquez ML, Kopatsis AD, Ouwehand AC, Forssten SD, Mukerji P, Caverly Rae JM, Dragan YP, Damewood JR, Tiihonen K, Ibarra A. Development of dietary soluble fibres by enzymatic synthesis and assessment of their digestibility in in vitro, animal and randomised clinical trial models. Int J Food Sci Nutr. 2017 Nov;68(7):849-864. doi: 10.1080/09637486.2017.1295027. Epub 2017 Mar 1. PMID 28276900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited through the Study site (Leatherhead Food Research, UK) volunteer database in September - October 2015.
Pre-assignment Details: 13 healthy volunteers were recruited, 12 volunteers were screened and one excluded (did not meet inclusion criteria).
Groups:
- Polydextrose First, Then Dextrose, Fibre1 and Fibre 2: Participant received study products at 4 visits, always diluted in 250 ml of water. Minimum washout period was 48 hours between consecutive visits. At first visit participant received 21.48 g Polydextrose Control, at second visit 23.89 g Dextrose Control, at third visit 22.17 g Dietary Fibre 1 and at fourth visit 21.48 g Dietary Fibre 2.
- Dextrose First, Then Fibre1, Fibre 2 and Polydextrose: Participant received study products at 4 visits, always diluted in 250 ml of water. Minimum washout period was 48 hours between consecutive visits. At first visit participant received 23.89 g Dextrose Control, at second visit 22.17 g Dietary Fibre 1, at third visit 21.48 g Dietary Fibre 2 and at fourth visit 21.48 g Polydextrose Control.
- Fibre1 First, Then Fibre 2, Polydextrose and Dextrose: Participant received study products at 4 visits, always diluted in 250 ml of water. Minimum washout period was 48 hours between consecutive visits. At first visit participant received 22.17 g Dietary Fibre 1, at second visit 21.48 g Dietary Fibre 2, at third visit 21.48 g Polydextrose Control and at fourth visit 23.89 g Dextrose Control.
- Fibre 2 First, Then Polydextrose, Dextrose and Fibre1: Participant received study products at 4 visits, always diluted in 250 ml of water. Minimum washout period was 48 hours between consecutive visits. At first visit participant received 21.48 g Dietary Fibre 2, at second visit 21.48 g Polydextrose Control, at third visit 23.89 g Dextrose Control and at fourth visit 22.17 g Dietary Fibre 1.
Period: First Intervention at Visit 1
Arm/Group | Polydextrose First, Then Dextrose, Fibre1 and Fibre 2 | Dextrose First, Then Fibre1, Fibre 2 and Polydextrose | Fibre1 First, Then Fibre 2, Polydextrose and Dextrose | Fibre 2 First, Then Polydextrose, Dextrose and Fibre1
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention at Visit 2
Arm/Group | Polydextrose First, Then Dextrose, Fibre1 and Fibre 2 | Dextrose First, Then Fibre1, Fibre 2 and Polydextrose | Fibre1 First, Then Fibre 2, Polydextrose and Dextrose | Fibre 2 First, Then Polydextrose, Dextrose and Fibre1
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention at Visit 3
Arm/Group | Polydextrose First, Then Dextrose, Fibre1 and Fibre 2 | Dextrose First, Then Fibre1, Fibre 2 and Polydextrose | Fibre1 First, Then Fibre 2, Polydextrose and Dextrose | Fibre 2 First, Then Polydextrose, Dextrose and Fibre1
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention at Visit 4
Arm/Group | Polydextrose First, Then Dextrose, Fibre1 and Fibre 2 | Dextrose First, Then Fibre1, Fibre 2 and Polydextrose | Fibre1 First, Then Fibre 2, Polydextrose and Dextrose | Fibre 2 First, Then Polydextrose, Dextrose and Fibre1
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received every study intervention in randomized order: Experimental Dietary Fibre 1 and 2, Polydextrose and Dextrose
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.09 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of IAUC (Incremental Area Under the Curve) in Blood Glucose Response
Time Frame: 0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes post dose
Population: Participants from whom full set of blood glucose measurements were available.
Measure: Mean (Standard Deviation); unit: min*mmol/L
Groups:
- Polydextrose Control: Polydextrose: 21.48 g of product diluted in 250 ml of water taken once orally.
Arm/Group | Experimental Dietary Fibre 1 | Experimental Dietary Fibre 2 | Polydextrose Control | Dextrose Control
Number analyzed (Participants) | 11 | 11 | 11 | 11
min*mmol/L | 127.45 (52.24) | 143.53 (52.11) | 19.27 (8.03) | 134.21 (59.00)

2. Secondary Outcome: Assessment of IAUC (Incremental Area Under the Curve) in Blood Insulin Response
Time Frame: 0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes post dose
Population: Participants from whom full set of blood insulin measurements were available.
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | Experimental Dietary Fibre 1 | Experimental Dietary Fibre 2 | Polydextrose | Dextrose Control
Number analyzed (Participants) | 9 | 9 | 9 | 9
min*mmol/L | 595.49 (151.72) | 640.94 (286.52) | 63.37 (55.81) | 687.13 (257.67)

ADVERSE EVENTS:
Arm/Group | Experimental Dietary Fibre 1 | Experimental Dietary Fibre 2 | Polydextrose Control | Dextrose Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 2/11 | 0/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Dietary Fibre 1 (N=11) | Experimental Dietary Fibre 2 (N=11) | Polydextrose Control (N=11) | Dextrose Control (N=11)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot release information without the sponsor's approval.